CLINICAL TRIAL: NCT00699946
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Perioperative Administration of Olanzapine to Prevent Postoperative Delirium in Joint Replacement Patients
Brief Title: Prophylactic Olanzapine Versus Placebo for Prevention of Postoperative Delirium After Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The New England Baptist Hospital (Other)
Responsible Party: Ken Larsen, Director, Pastoral Care/Psychology, New England Baptist Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7381*KELLY
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Delirium
Keywords: delirium, atypical antipsychotics, olanzapine, orthopedic
MeSH Terms: conditions — Delirium | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: olanzapine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — 5 mg preoperative and 5mg postoperative prior to discharge to inpatient nursing floor
  Other Names: Zyprexa
  Arms: 1
Drug: placebo — placebo administered preoperatively and postoperatively prior to discharge to inpatient nursing floor
  Arms: 2

SUMMARY:
In this study we wanted to determine if perioperative administration of olanzapine prior to knee or hip replacement surgery in high risk patients would prevent the onset of postoperative delirium.

DETAILED DESCRIPTION:
Postoperative delirium is a serious and common (20% to 60%) complication in orthopedic surgery patients. In this study we investigate whether prophylactic administration of olanzapine can prevent delirium from occurring after knee or hip replacement in high-risk patients > 65 years of age. This is a randomized, double-blind, single center, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* High risk for delirium age > 65 history of delirium medical comorbidities ability to give informed consent

Exclusion Criteria:

* Dementia Alcohol abuse Current use of an antipsychotic Allergy to olanzapine

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 495 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
incidence of delirium | days in hospital

SECONDARY OUTCOMES:
Complications, length of stay, hospital costs | days

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kelly, MD, Principal Investigator — New England Baptist Hospital
Locations (1):
- New England Baptist Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Larsen KA, Kelly SE, Stern TA, Bode RH Jr, Price LL, Hunter DJ, Gulczynski D, Bierbaum BE, Sweeney GA, Hoikala KA, Cotter JJ, Potter AW. Administration of olanzapine to prevent postoperative delirium in elderly joint-replacement patients: a randomized, controlled trial. Psychosomatics. 2010 Sep-Oct;51(5):409-18. doi: 10.1176/appi.psy.51.5.409. PMID 20833940